CLINICAL TRIAL: NCT02969070
Title: Randomized Trial to Evaluate the Effects of Two Different Nutraceutical Therapies on Endothelial Function, Platelet Aggregation, and Coronary Flow Reserve in Hypercholesterolemic Patients at Moderate Cardiovascular Risk
Brief Title: Effects of Nutraceutical Therapies on Endothelial Function, Platelet Aggregation, and Coronary Flow Reserve
Acronym: NUTRENDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Bruno Trimarco, Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FedericoIIU 259/16
Record Dates: First submitted 2016-11-13; First posted 2016-11-21 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Hypercholesterolemia; Endothelial Dysfunction
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LopiGLIK™ group (Active Comparator): 4 weeks of LopiGLIK™ therapy 1 capsule/day
  Interventions: Dietary Supplement: LopiGLIK™ therapy
- Armolipid Plus group (Active Comparator): 4 weeks of Armolipid Plus therapy 1 capsule/day
  Interventions: Dietary Supplement: Armolipid Plus® therapy

INTERVENTIONS:
Dietary Supplement: LopiGLIK™ therapy — 4 weeks of LopiGLIK™ therapy 1 capsule/day
  Arms: LopiGLIK™ group
Dietary Supplement: Armolipid Plus® therapy — 4 weeks of Armolipid Plus® therapy 1 capsule/day
  Arms: Armolipid Plus group

SUMMARY:
Hypercholesterolemia is considered one of the most important cardiovascular risk factors. Cardiovascular prevention include a class I indication to statins in addition to non-pharmacologic intervention and prevention strategies in patients deemed to be 'high risk'. Along with non-pharmacologic intervention and prevention strategies, newer approaches to reduce cholesterol blood levels currently include nutraceuticals, which are compounds derived from foods with cholesterol lowering actions. However, it remains unclear if nutraceuticals yield additive positive effects other than cholesterol lowering. In particular, there is evidence that Berberine has cardiovascular protective effects and that, in vitro, Morus Alba, mulberry fruit, modulates platelet function by inhibiting platelet activation, thromboxane formation, serotonin secretion, aggregation and thrombus formation. Furthermore, Morus Alba exerts an α-glucosidase inhibitory and antioxidant activity in vitro, which may reduce postprandial glucose peak, thus improving HbA1c concentration. Accordingly, we designated a study to evaluate the effects of two commercially available nutraceutical combined pills [LopiGLIK™, Akademy Pharma, 1 capsule/day containing red yeast rice 220 mg (at least 3,3 mg of Monacolin K) + Berberine 531,25 mg + Morus Alba 200 mg (at least 4 mg of Deoxynojirimycin) vs. Armolipid Plus®, Meda Pharma, 1 capsule/day containing Berberis aristata d.e. 588 mg (equivalent to Berberine chloride 500 mg) + Red yeast rice 200 mg (equivalent to Monacolin K 3 mg) + Policosanol 10 mg + Folic acid 0.2 mg + Coenzyme Q10 2.0 mg + Astaxanthin 0.5 mg] on lipid and metabolic profile, platelet aggregation, endothelial function and coronary flow reserve (CFR). For this purpose patients with hypercholesterolemia not requiring statins or statin intolerant at moderate cardiovascular risk will be subjected at day 0 and at day 28, after 4 weeks of therapy, to blood sampling to evaluate lipid and metabolic profile, peripheral arterial tonometry (EndoPAT), platelet aggregation tests with light transmission aggregometry (LTA), nitric oxide (NO) release, endothelial nitric oxide synthase (eNOS) phosphorylation on platelets. Only for CFR, patients will be further evaluated also after two hours from the administration of the first dose of nutraceutical combined pill. Patients will be randomly assigned to receive therapy with LopiGLIK™ or with Armolipid Plus®.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) are the principal cause of death worldwide. Primary prevention of cardiovascular disease by identifying and treating at-risk individuals remains a major public-health priority. According to guidelines, the main approach is a healthy life-style, assisted by pharmaco-therapy. Hypercholesterolemia is considered one of the most important cardiovascular risk factors. Cardiovascular prevention include a class I indication to statins in addition to non-pharmacologic intervention and prevention strategies in patients deemed to be 'high risk'. In the real world, however, statin treatment is often discontinued due to side effects. In addition, statins are not indicated in those subjects deemed to be 'low risk', in whom only non-pharmacologic intervention and prevention strategies are currently prescribed. Along with non-pharmacologic intervention and prevention strategies, newer approaches to reduce cholesterol blood levels currently include nutraceuticals, which are compounds derived from foods with cholesterol lowering actions. However, it remains unclear if nutraceuticals yield additive positive effects other than cholesterol lowering. In particular, there is evidence that Berberine has cardiovascular protective effects and that, in vitro, Morus Alba, mulberry fruit, modulates platelet function by inhibiting platelet activation, thromboxane formation, serotonin secretion, aggregation and thrombus formation. Furthermore, Morus Alba exerts an α-glucosidase inhibitory and antioxidant activity in vitro, which may reduce postprandial glucose peak, thus improving HbA1c concentration. Accordingly, we designated a study to evaluate the effects of two commercially available nutraceutical combined pills [LopiGLIK™, Akademy Pharma, 1 capsule/day containing red yeast rice 220 mg (at least 3,3 mg of Monacolin K) + Berberine 531,25 mg + Morus Alba 200 mg (at least 4 mg of Deoxynojirimycin) vs. Armolipid Plus®, Meda Pharma, 1 capsule/day containing Berberis aristata d.e. 588 mg (equivalent to Berberine chloride 500 mg) + Red yeast rice 200 mg (equivalent to Monacolin K 3 mg) + Policosanol 10 mg + Folic acid 0.2 mg + Coenzyme Q10 2.0 mg + Astaxanthin 0.5 mg] on lipid and metabolic profile, platelet aggregation, endothelial function and coronary flow reserve (CFR). For this purpose patients with hypercholesterolemia not requiring statins or statin intolerant at moderate cardiovascular risk will be subjected at day 0 and at day 28, after 4 weeks of therapy, to blood sampling to evaluate lipid and metabolic profile, peripheral arterial tonometry (EndoPAT), platelet aggregation tests with light transmission aggregometry (LTA), NO release, eNOS phosphorylation on platelets. Only for CFR, patients will be further evaluated also after two hours from the administration of the first dose of nutraceutical combined pill. Patients will be randomly assigned to receive therapy with LopiGLIK™ or with Armolipid Plus®.

STUDY DESIGN

Study procedure For study enrolment, all subjects will undergo a screening to determine the criteria for inclusion / exclusion in the study. Eligible patients will receive an information sheet that will give a preview to the family and to General Practitioner, and, if accept to participate, they must sign a written informed consent.

The information collected for each subject, regarding suitability to the study, will be retained and stored by Investigators.

Condition Outcomes Intervention

Patients with hypercholesterolemia and moderate cardiovascular risk according to current European Society of Cardiology (ESC) guidelines Device: Peripheral arterial tonometry (EndoPAT) Device: Platelet aggregation with LTA Platelet isolation for measurement of eNOS phosphorylation Device: colorDoppler echocardiography at rest and after cold pressure test for CFR evaluation 4 weeks of LopiGLIK™ therapy

1 capsule/day or 4 weeks of Armolipid Plus® therapy

1 capsule/day

Study Type: Interventional

Study plan:

* 30 patients will be evaluated at day 0 (anamnesis, cardiovascular risk factors, medications, EndoPAT + CFR + blood sample (1 yellow tube for biochemistry + 6 light blue tubes for platelet function)
* Patients will be randomly assigned to treatment for 4 weeks with 1 capsule/day of LopiGLIK™ containing red yeast rice 220 mg + Berberine 531,25 mg + Morus Alba 200 mg or with 1 capsule/day of Armolipid Plus® containing Berberis aristata d.e. 588 mg (equivalent to Berberine chloride 500 mg) + Red yeast rice 200 mg (equivalent to Monacolin K 3 mg) + Policosanol 10 mg + Folic acid 0.2 mg + Coenzyme Q10 2.0 mg + Astaxanthin 0.5 mg
* Re-evaluation at day 28 of all tests performed at day 0

Primary Outcome Measures:

• Effects on endothelial function as evaluated by Reactive Hyperemia Index (RHI)

Secondary Outcome Measures:

* Evaluation of treatment tolerability (as evaluated by a specific questionnaire)
* Reasons for treatment discontinuation
* Effects on lipid profile (total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides) and metabolic indexes (glucose levels, insulin plasma levels, insulin sensitivity index (HOMA index)
* Effects on platelet aggregation as evaluated by LTA
* Effects on coronary flow reserve (CFR) as evaluated by echocardiocolorDoppler visualization of coronary flow in the distal left anterior descending artery at rest and after cold pressure test (CPT).

STUDY POPULATION

30 patients will be enrolled (15 in each treatment group).

METHODS

Endothelial function Endothelial function will be assessed with the flow-mediated dilation test (FMD) by digital pulse amplitude, using a fingertip PAT as previously described [Gargiulo P, et al. Int J Cardiol 2013]. The system (Itamar Medical Ltd., Caesarea, Israel) consists of a finger probe to assess digital volume changes accompanying pulse waves. All subjects included in the study were maintained without smoking, alcohol or caffeine from the night before the evaluation. Reactive hyperaemia was measured as a PAT reactive hyperaemic index (RHI) calculated as the ratio of the average amplitude of the PAT signal over a 1-min time interval starting 1-min after cuff deflation divided by the average amplitude of the PAT signal of a 3.5-min time period before cuff inflation (baseline) and normalized to the RHI of the control arm. Endothelial dysfunction was defined as a RHI <1.68 calculated by the mean value minus 2 standard deviations of 20 healthy asymptomatic control individuals without history of cardiovascular disease and without major cardiovascular risk factors as previously described.

Platelet function Platelet aggregation will be measured by light transmission aggregometry (LTA) using a dual channel lumi-aggregometer (model 700; Chrono-Log). Platelets will be prepared according to a standard procedure. Briefly, platelet-rich plasma (PRP) will be prepared from blood that was drawn by venipuncture into 3.8% trisodium citrate (w/v) Vacutainer Blood Collection Tubes. PRP will be obtained by centrifugation of blood at 250 g at 25°C for 15 minutes. Platelet-poor plasma (PPP) will be obtained by centrifugation of the rest of the blood at 1400 g at 25°C for 10 minutes.

Platelet aggregation will be monitored at 37°C with constant stirring (1200 rpm) and measured as the increase in light transmission for 10 minutes, with the addition of adenosine diphosphate (ADP) 10 μmol/L, collagen 2 μg/ml and arachidonic acid 1 0,5 millimole (mM) as a proaggregatory stimulus. All measurements will be obtained within 2 hours of sample collection, and results will be reported as percentage maximum aggregation. Some experiments will be performed in platelet pre-treated with insulin (15 microIU/mL) for 30 minutes at 37°C. After stimulation, 3 ml of platelet suspension will be centrifuged for 15 minutes at 3000 and the platelet pellet obtained will be used for the measurement of eNOS phosphorylation and NO levels.

Coronary flow reserve Standard Doppler echocardiography will be performed using a Vivid Seven machine (GE, Horten, Norway) in the morning after an overnight fast of 12-14 h; subjects will be instructed to avoid all coffee-containing drinks and theophylline containing medications, and to abstain from smoking and heavy exercise from 24 h before the study. The color Doppler visualization of coronary flow in the distal left anterior descending artery will be obtained with a 5 megahertz (MHz) shallow-focus phased-array transducer. Doppler sample volume will be placed on the color signal of the left anterior descending artery, and the spectral pulsed Doppler signal will be recorded to look for the characteristic biphasic flow pattern with a larger diastolic and a smaller systolic component both at rest and after cold pressure test (CPT). Coronary diastolic peak flow velocities (cm/s) as well as heart rate and BP will be measured at rest and soon after CPT, corresponding to maximal hyperemia. CFR will be calculated as the ratio of hyperemic-to-resting diastolic peak velocities. The CPT will be performed according to a standardized protocol, by placing the subject's hand and distal part of the forearm in an ice water slurry for 3 min. The highest three spectral Doppler signals will be averaged for each parameter. CFR will be evaluated at baseline, 2 hours after administration of the first nutraceutical combined pill, and after 28 days of therapy.

All images will be recorded on local archives and analyzed off-line by two observers who will be blinded to the clinical characteristics of the patients.

Sample size calculation Assuming that the standard deviation of the differences in Endo-PAT indices for the 2 test days would be 0.5 and that we would want to detect a true difference in means >0.5 with a paired t test conducted at the 0.05 level of significance, we determined that a sample of 30 subjects (15 for each group) would provide 80% power.

Composition and supply of the nutraceutical treatments Capsules of LopiGLIK™ (containing red yeast rice 220 mg + Berberine 531,25 mg + Morus Alba 200 mg) and of Armolipid Plus® (containing Berberis aristata d.e. 588 mg (equivalent to Berberine chloride 500 mg) + Red yeast rice 200 mg (equivalent to Monacolin K 3 mg) + Policosanol 10 mg + Folic acid 0.2 mg + Coenzyme Q10 2.0 mg + Astaxanthin 0.5 mg) will be provided free of charge by Akademy Pharma and Meda Pharma, respectively.

Treatment duration All patients will be treated for a period of 4 weeks.

Data Results of the study will be communicated to all participant at the study end.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old
2. Patients with hypercholesterolemia and moderate cardiovascular risk according to current ESC guidelines (risk of fatal cardiovascular event of 1-9% at 10 years according to SCORE risk charts of low-risk populations)
3. Patients giving written Informed Consent.

Exclusion Criteria:

1. Statin treatment indication
2. Previous cardiovascular event
3. Diabetes mellitus
4. Creatinine Clearance <60ml/min/1.73mm2
5. Moderate to severe anemia Hb < 10mg/dl
6. Platelet count >600 x 103/mm3 o <150 x 103/mm3 o hematocrit (HCT) >50% o <25%

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-11; Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Effects on endothelial function as evaluated by Reactive Hyperemia Index (RHI) | 28 days

SECONDARY OUTCOMES:
Evaluation of treatment tolerability | 28 days
  Self reporting questionnaire
Reasons for treatment discontinuation | 28 days
  Self reporting questionnaire
Effects on lipid profile (total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides) | 28 days
  mg/dL
Effects on metabolic indexes (glucose levels) | 28 days
  mg/dL
Effects on metabolic indexes [insulin plasma levels and insulin sensitivity index (HOMA index)] | 28 days
  microIU/mL
Effects on platelet aggregation as evaluated by light transmission aggregometry (LTA) | 28 days
Effects on coronary flow reserve (CFR) as evaluated by echocardiocolorDoppler visualization of coronary flow in the distal left anterior descending artery at rest and after cold pressure test (CPT) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Trimarco, MD, Principal Investigator — Federico II University
Locations (1):
- University of Naples "Federico II", Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Piepoli MF, Hoes AW, Agewall S, Albus C, Brotons C, Catapano AL, Cooney MT, Corra U, Cosyns B, Deaton C, Graham I, Hall MS, Hobbs FDR, Lochen ML, Lollgen H, Marques-Vidal P, Perk J, Prescott E, Redon J, Richter DJ, Sattar N, Smulders Y, Tiberi M, van der Worp HB, van Dis I, Verschuren WMM, Binno S; ESC Scientific Document Group. 2016 European Guidelines on cardiovascular disease prevention in clinical practice: The Sixth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of 10 societies and by invited experts)Developed with the special contribution of the European Association for Cardiovascular Prevention & Rehabilitation (EACPR). Eur Heart J. 2016 Aug 1;37(29):2315-2381. doi: 10.1093/eurheartj/ehw106. Epub 2016 May 23. No abstract available. PMID 27222591
- [Background] Trimarco V, Izzo R, Stabile E, Rozza F, Santoro M, Manzi MV, Serino F, Schiattarella GG, Esposito G, Trimarco B. Effects of a new combination of nutraceuticals with Morus alba on lipid profile, insulin sensitivity and endotelial function in dyslipidemic subjects. A cross-over, randomized, double-blind trial. High Blood Press Cardiovasc Prev. 2015 Jun;22(2):149-54. doi: 10.1007/s40292-015-0087-2. Epub 2015 Apr 14. PMID 25870124
- [Background] Carrizzo A, Ambrosio M, Damato A, Madonna M, Storto M, Capocci L, Campiglia P, Sommella E, Trimarco V, Rozza F, Izzo R, Puca AA, Vecchione C. Morus alba extract modulates blood pressure homeostasis through eNOS signaling. Mol Nutr Food Res. 2016 Oct;60(10):2304-2311. doi: 10.1002/mnfr.201600233. Epub 2016 Jun 27. PMID 27234065
- [Background] Gargiulo P, Marciano C, Savarese G, D'Amore C, Paolillo S, Esposito G, Santomauro M, Marsico F, Ruggiero D, Scala O, Marzano A, Cecere M, Casaretti L, Perrone Filardi P. Endothelial dysfunction in type 2 diabetic patients with normal coronary arteries: a digital reactive hyperemia study. Int J Cardiol. 2013 Apr 30;165(1):67-71. doi: 10.1016/j.ijcard.2011.07.076. Epub 2011 Aug 17. PMID 21851998
- [Background] Marciano C, Galderisi M, Gargiulo P, Acampa W, D'Amore C, Esposito R, Capasso E, Savarese G, Casaretti L, Lo Iudice F, Esposito G, Rengo G, Leosco D, Cuocolo A, Perrone-Filardi P. Effects of type 2 diabetes mellitus on coronary microvascular function and myocardial perfusion in patients without obstructive coronary artery disease. Eur J Nucl Med Mol Imaging. 2012 Jul;39(7):1199-206. doi: 10.1007/s00259-012-2117-9. Epub 2012 Apr 12. PMID 22526959
- [Derived] Esposito R, Sorrentino R, Giugliano G, Avvedimento M, Paolillo R, Santoro C, Scalamogna M, Esposito M, Ilardi F, Rozza F, Esposito G, Galderisi M, Trimarco V. Different age-independent effects of nutraceutical combinations on endothelium-mediated coronary flow reserve. Immun Ageing. 2018 Nov 22;15:30. doi: 10.1186/s12979-018-0138-3. eCollection 2018. PMID 30479642